CLINICAL TRIAL: NCT02690818
Title: Promoting Adherence to Treatment for Latent TB Infection Through Mobile Phone Text Messaging
Brief Title: Promoting Adherence to Treatment for Latent TB Infection Through Text Messaging
Acronym: TXT4MED
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Arizona (Other)
Collaborators: Pima County Health Department (Unknown); American Lung Association (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: TXT4MED
Record Dates: First submitted 2016-01-05; First posted 2016-02-24 (Estimated); Last update posted 2019-04-23 (Actual); Status verified 2019-04

CONDITIONS: Latent Tuberculosis
Keywords: Tuberculosis; Latent Tuberculosis; Texting; Adherence; Medication
MeSH Terms: conditions — Latent Tuberculosis; Tuberculosis

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Behavioral intervention arm (Experimental): Regularly scheduled medication reminder text messages
  Daily LTBI text messages without the option to text back. The messages will read, "This is a reminder to take your medication."
  Standard of care: Monthly reminder call and clinic visit
  Interventions: Behavioral: Regularly scheduled LTBI medication reminder text messages
- Control group receiving standard care (No Intervention): Standard of care: Monthly reminder call and clinic visit

INTERVENTIONS:
Behavioral: Regularly scheduled LTBI medication reminder text messages — Regularly scheduled medication reminder text messages Daily LTBI text messages without the option to text back. The messages will read, "This is a reminder to take your medication."
  Arms: Behavioral intervention arm

SUMMARY:
The purpose of this pilot study is to determine whether regularly scheduled medication reminder text messages (SMS) are effective in increasing latent tuberculosis infection (LTBI) treatment completion.

DETAILED DESCRIPTION:
We aim to determine the feasibility and acceptability of text reminders for improving adherence in latent TB patients. Specific objectives of the current study are to: 1) Assess the feasibility of the intervention as indicated by participant recruitment and retention and; 2) Evaluate the acceptability of the intervention, as indicated by intervention adherence, outcome measurement rates, and feedback from participants.

Data will be used to design a definitive trial which will test the hypothesis that the intervention will improve medication adherence, as measured through an increase in treatment completion rates, and result in higher self-reported medication adherence, fewer missed appointments and doses, and a shorter course of treatment.

ELIGIBILITY:
Inclusion Criteria:

* Consent to the study
* Own a mobile phone which operates on a telecom provider supported by our SMS platform
* Initiating or actively receiving treatment for LTBI at the Pima County TB Clinic in Tucson, AZ
* Prescribed self-administered therapy
* Report not having prior or current active TB disease
* Know how to and are able to receive SMS messages
* At least 18 years of age

Exclusion Criteria:

* Do not meet inclusion criteria
* Do not consent to study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2016-04; Primary Completion 2018-09-26 (Actual); Study Completion 2018-09-26 (Actual)

PRIMARY OUTCOMES:
Recruitment | Ongoing
  How many approached by clinic, how many referred, how many study eligible, how many consented; why ineligible or refused; how long to recruit each patient

SECONDARY OUTCOMES:
Retention | Ongoing
  How many drop out at each monthly time point, who and why
Perceptions of Intervention through a questionnaire | Once, up to 12 months post-treatment
  Perceptions and opinions (if the intervention was helpful, non-helpful, effectiveness) in the intervention arm will be assessed after the study follow-up through a questionnaire of a subset of enrolled individuals at the completion of the participant's treatment (up to 12 months post-treatment initiation).

CONTACTS AND LOCATIONS:
Overall Officials: Eyal Oren, PhD, Principal Investigator — University of Arizona
Locations (1):
- Pima County Health Department, Tucson, Arizona, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Oren E, Bell ML, Garcia F, Perez-Velez C, Gerald LB. Promoting adherence to treatment for latent TB infection through mobile phone text messaging: study protocol for a pilot randomized controlled trial. Pilot Feasibility Stud. 2017 Mar 13;3:15. doi: 10.1186/s40814-017-0128-9. eCollection 2017. PMID 28293431